CLINICAL TRIAL: NCT00744913
Title: Randomized, Controlled Open-Label Study of Nicotine Replacement Therapy in Pregnancy
Brief Title: Study of Nicotine Replacement Therapy in Pregnancy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Discontinued due to difficulty in recruitment
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Gideon Koren, Director of MotherRisk Program, Clinical Pharmacology and Toxicology, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000010740
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Smoking Cessation
Keywords: Pregnancy; Women; Nicotine replacement therapy; Smoking cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Nicoderm patches
- 2 (Active Comparator)
  Interventions: Other: Counselling

INTERVENTIONS:
Drug: Nicoderm patches — Women in this group will receive standard counselling and NRT (Nicoderm patches) starting with a dose of 14 mg/day that can be increased to 21 mg/day based on response (smoking cessation) and potential side effects
  Arms: 1
Other: Counselling — Women in this arm of the study will receive standard counseling only.
  Arms: 2

SUMMARY:
The overall objective of this study is to assess the effectiveness of NRT (Nicoderm patches) plus counselling treatment in women in the second and third trimester of pregnancy.

DETAILED DESCRIPTION:
Smoking during pregnancy is a major public health issue, causing miscarriages, prematurity, intrauterine growth retardation, stillbirth, and the Sudden Infant Death Syndrome (SIDS). It is estimated that 25-40% of pregnant smokers try to stop smoking on their own upon learning that they are pregnant. While pregnancy is often a strong motivator for smoking cessation, many nicotine-dependent women cannot quit smoking. The most important factor underlying the inability to quit smoking is strong dependence on a certain level nicotine, which is unique in every individual.

Several publications have shown that the use of the nicotine patch during the second and third trimesters is not associated with maternal or fetal compromise. More importantly, nicotine replacement therapy (NRT) during pregnancy exposes the fetus to lower levels of nicotine than smoking cigarettes does and, moreover, eliminates exposure to numerous other toxic substances.

Presently, counselling is the standard mode of treatment for the pregnant patients willing to quit smoking. Since pharmacologic smoking cessation therapies have been shown to increase significantly up to doubling a successful quitting rate when used in adjunction to brief physician counselling, the use of an appropriate dose of such agents is essential.

ELIGIBILITY:
Inclusion Criteria:

* Women who smoke
* Pregnant women after 12 weeks gestation, confirmed by ultrasound
* On the day of the recruitment, women will be at least 18 years old and no older than 40 years old
* Agree to sign consent form and participate in all aspects of the follow-up

Exclusion Criteria:

* Women who refuse to participate in the study/sign a written consent
* Women with insufficient English language skills to understand the questionnaires and assessment material
* Women with multiple pregnancy
* Women with confirmed cardiac pathology
* Women who receive concurrent treatment with Bupropion
* Congenital malformations visualized by ultrasound
* Objection from the physician caring for the woman to her participation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2010-02 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
To assess the effectiveness of NRT (Nicoderm patches) at doses of 14 mg/day or 21 mg/day plus counselling treatment | 6 months

SECONDARY OUTCOMES:
To compare the effectiveness of counseling and NRT at doses of 14 mg/day or 21 mg/day with counselling alone. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gideon Koren, MD, Principal Investigator — The Hospital for Sick Children